CLINICAL TRIAL: NCT06102811
Title: Low Concentration Local Anesthesia Fascia Iliaca Block for Total Hip Arthroplasty
Acronym: HALF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Hermann dos Santos Fernandes, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22-0206-A
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Concentration Local Anesthetic Fascia Iliaca Compartment Block (Experimental): Patients will be submitted to a Suprainguinal Fascia Iliaca Block with low concentration local anesthetic (Ropivacaine 0.075%)
  Interventions: Other: Low Concentration Local Anesthetic Fascia Iliaca Compartment Block
- High Concentration Local Anesthetic Fascia Iliaca Compartment Block (Active Comparator): Patients will be submitted to a Suprainguinal Fascia Iliaca Block with high concentration local anesthetic (Ropivacaine 0.25%)
  Interventions: Other: High Concentration Local Anesthetic Fascia Iliaca Compartment Block

INTERVENTIONS:
Other: Low Concentration Local Anesthetic Fascia Iliaca Compartment Block — Fascia iliaca block with Ropivacaine 0.075% (50 mL)
  Arms: Low Concentration Local Anesthetic Fascia Iliaca Compartment Block
Other: High Concentration Local Anesthetic Fascia Iliaca Compartment Block — Fascia iliaca block with Ropivacaine 0.25% (50 mL)
  Arms: High Concentration Local Anesthetic Fascia Iliaca Compartment Block

SUMMARY:
Fascia iliaca compartment block (FICB) is a documented option for postoperative analgesia for total hip arthroplasty (THA) surgery. FICB is demonstrated to be effective in terms of analgesia and opioid requirements decrease, however it causes quadriceps motor weakness. Current available motor sparing techniques are not as effective as FICB for analgesia. Low concentration local anesthetics (LCLA) are used with excellent results for pain control with no or minimum motor block effect, in other scenarios (highlighted in obstetric anesthesia) and techniques (epidural anesthesia, for instance). This study proposes that LCLA-FICB can offer the benefit of peripheral nerve blocks mediated analgesia, while at the same time avoiding motor blockade and muscle weakness. The investigators hypothesize that LCLA-FICB, when compared to conventional high concentration local anesthetics (HCLA) FICB, provides similar postoperative analgesia in the first 24 hours following primary THA, while at the same time preserving quadriceps muscle group strength.

DETAILED DESCRIPTION:
Significance There are no published prospective randomized controlled trials evaluating LCLA blocks for THA. As THA is the second most frequent type of surgery requiring hospitalization, and has the prediction to increase its incidence for the next years, there is significant importance in investigations about interventions which may improve its recovery in an outpatient regime. A postoperative analgesic technique that offers better pain control, has less adverse effects, reduces the opioid analgesia requirement and is safer, may have additional impact on decreasing health care costs, and may lead to an enhanced recovery and better quality of life for THA patients.

Objectives The primary objective will be to evaluate efficacy of LCLA-FICB in comparison to HCLA-FICB for patients undergoing primary THA, in terms of pain scores and opioid consumption.

The secondary objective is to assess postoperative opioid related side effects and ipsilateral quadriceps weakness between those two postoperative analgesia techniques.

Hypothesis The LCLA-FICB, in comparison to HCLA-FICB, provides non-inferior postoperative analgesia in the first 24 hours following primary THA, while at the same time preserving quadriceps muscle group strength.

Methods Study type This will be a randomized controlled prospective trial, blinded for patient and evaluator, in patients undergoing primary THA at Sinai Health. After Hospital's Ethics in Research Board approval, the recruitment will begin. Patients will be assessed about their eligibility for participating and after plain clear information about the study interventions they will or will not authorize their inclusion and data collection, through the signature of a written consent.

Perioperative management and interventions The subjects will have their surgeries booked in advance and they will be submitted to the pre anesthesia consult at the Pre-Admission Unit (PAU) a few days before the surgery. The study proposal will be explained to the patients on that occasion and they will receive the consent form, with the information about the study, that they will bring home to review. They will have the time between the pre anesthesia assessment and the surgery (at least 24 hours) to review and consent to the study.

Patients will be randomized to one of the two groups using a computer-generated random numbers table. The randomization will be done before the beginning of the study and will define which study number is going to be managed as intervention group (LCLA-FICB) or control group (HCLA-FICB). Each patient will receive a study number following the order of their entrance on the study and that number will be already linked for one of the two groups. Closed envelopes will be prepared ahead of time and each of them will have the name of the group related to its study number. Once the patient is included, the research coordinator will check inside the envelope which group the patient is randomized to, in order to prepare the solution for the FICB (LCLA or HCLA). A list with the study numbers and the randomization will be kept by the research coordinator, under password protection, and will be shared with other researches only after all data collection is finished. The patient, the research assistant, the professional who performs the postoperative assessments and the professional providing anesthesia care to the patient will be blinded to which group each patient is randomized to.

All patients will receive the same perioperative management. Patients will initially be brought to a dedicated block room where a safety checklist will be performed by the block room team. Standard Canadian Anesthesia Society monitoring will be provided. Mild sedation with Midazolam 0.5-2mg and Fentanyl 25-150mcg might be administered for anxiolysis and analgesia. After proper cleaning of the ipsilateral hip area, under sterile technique and ultrasound guidance (Sonosite Edge II ultrasound machine), a supra-inguinal FICB will be performed21. Patients in the LCLA-FICB group will receive a block with 50 ml of Ropivacaine 0.075 % with epinephrine 1:200,000. Patients in the control group (HCLA-FICB) will receive a supra-inguinal FICB block with 50 ml of Ropivacaine 0.25% with epinephrine 1:200,000 (concentration of local anesthetics used routinely for this PNB).

After the FICB block is performed, all patients will receive standard spinal anesthesia using Mepivacaine 2% x 3.5 ml with fentanyl 15 mcg and preservative free morphine 100 mcg. All intraoperative opioids administered will be recorded. In the intra-operative period, each patient will receive IV Cefazolin 2-3 g, Tranexamic acid 20 mg/kg, Dexamethasone 0.1 mg/kg, and Ondansetron 4 mg.

Standard oral analgesic scheme will be prescribed to every patient (Acetaminophen 650 - 1000 mg QID, Celecoxib 100 - 200 mg BID, Hydromorphone 1 - 2 mg PRN Q2Hs, Hydromorphone 0.2 - 0.4 mg IV PRN Q1H).

Outcomes Patients will be assessed at 1-2h before surgery for demographic information (age, weight, height, body mass index, gender, ASA functional status) and baseline pain scores and average opioid consumption.

After the surgery, patients will be assessed in person, by a research team member, blinded to which group the patient was randomized to, on 4, 8, 24 and 48 hours after the spinal anesthesia moment, as following:

* 4 hours time point: pain scores, quadriceps muscle weakness, sensitive dermatomes, nerve block related complications, opioid consumption;
* 8 hours time point: pain scores, quadriceps muscle weakness, sensitive dermatomes, nerve block related complications;
* 24 hours time point: pain scores, quadriceps muscle weakness, sensitive dermatomes, nerve block related complications, opioid consumption;
* 48 hours time point: pain scores, quadriceps muscle weakness, sensitive dermatomes, nerve block related complications, opioid consumption.

The primary end point of the study is the degree of muscle weakness on 4 hours after surgery.. Secondary outcome parameters will include the following: total opioid consumption at 48 hours, pain scores, , dermatomes sensation impairment, nerve block related complicaitonsand hospital length of stay.

Pain will be measured using the numerical rating scale (NRS) for pain (0 = no pain at all, 10 = worst pain). For the 4- and 8-hours assessments, the patients will be asked to rate their lowest and highest pain scores for the last 4 and 8 hours. From the rest of the moments, they will be asked to rate their pain at rest and at movement (from sitting position to standing up). Opioid usage will be measure in oral morphine equivalent doses. Quadriceps weakness will be evaluated using the Muscle Strength Grading (Oxford Scale), by a member of the research team22: 0 - no muscle activation; 1 - trace muscle activation, such as a twitch, without achieving full range of motion; 2 - muscle activation with gravity eliminated, achieving full range of motion; 3 - muscle activation against gravity, full range of motion; 4 - muscle activation against some resistance, full range of motion; 5 - muscle activation against examiner's full resistance, full range of motion.

The dermatome sensibility assessment will be done by asking about how intense is the patient's sensation to an ice pack put on their anterior, medial or lateral aspect of the thigh, in comparison to the opposite side. If the could sensation is less intense than the opposite side, that nerve territory will be considered blocked to the ice sensation.

The potential complications related to the nerve block to be interrogated are: ipsilateral lower limb weakness, occurrence of fall, infection signs (redness, purulent secretion, local hyperthermia), pruritus sensation, burning sensation, tingling sensation, electrical shock sensation, symptoms or signs of LAST (any of the following: numbness on tongue and lips, diplopia, tinnitus, metal taste on mouth, seizure).

Sample size The sample size was calculated based on previous study that compared supra-inguinal FICB versus LAI, in 60 patients undergoing elective THA23. They found no difference between the groups for opioid consumption on the first 24h after the surgery, however the group FICB had higher occurrence of quadriceps muscle weakness on the first six hours after surgery. That study can be considered as comparing a muscle weakness associated technique (FICB) with a technique not associated with muscle weakness (LAI), which found a significant difference for quadriceps weakness incidence in a sample of 60 patients. Translating the same numbers for a similar study evaluating local anesthetic concentration and the occurrence of motor block (motor sparing concentration versus a non-sparing concentration), the investigators plan to include 30 patients per group.

Study data analysis Normal distributed variables values will be presented and analyzed as mean values ± standard deviation (SD). Non-normal distributed variables values will be presented and analyzed as median and minimum and maximum values. Qualitative variables will be presented as frequency of occurrence. Statistical test to be performed might be: t-Student, Kruskal-Wallis and Chi-square.. Study data will be collected and managed using a password protected Microsoft Excel sheet (Microsoft Corporation, 2018). Statistical software will be used for analysis: SPSS 13.0 for Windows (SPSS Inc, Chicago, IL, USA) and GraphPad Prism Version 4.00 for Windows (GraphPad Software, San Diego, CA, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary THA in the inpatient setting.
* Non-pregnant patients older than 21 years of age.
* Patients with American Society of Anesthesiologists (ASA) physical status I-IV.
* No alcohol or drug dependency.

Exclusion Criteria:

* Patients undergoing outpatient THA.
* Chronic opioid use of 30 mg or more of oral morphine equivalent, per day, for the last 2 consecutive weeks.
* Contraindications for nerve block placement (severe anatomic abnormalities, local or systemic infection).
* Contraindications for any of the standardized medications used for the study (Mepivacaine, Fentanyl, Dexamethasone, Ondansetron, Acetaminophen, Celecoxib, Hydromorphone).
* Not submitted to the standardized spinal anesthesia technique.
* Need to conversion to general anesthesia after the start of the surgery.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Quadriceps muscle strenght | 4 hours after spinal anesthesia
  Intensity of quadriceps strength: Muscle Strength Grading (Oxford Scale): 0 - no muscle activation; 1 - trace muscle activation, such as a twitch, without achieving full range of motion; 2 - muscle activation with gravity eliminated, achieving full range of motion; 3 - muscle activation against gravity, full range of motion; 4 - muscle activation against some resistance, full range of motion; 5 - muscle activation against examiner's full resistance, full range of motion.

SECONDARY OUTCOMES:
Pain scores | 24 hours after spinal anesthesia
  Numerical verbal scale (0 = no pain at all, 10 = worst pain)
Opioid consumption | 24 hours after spinal anesthesia
  Amount of opioids (in oral morphine equivalents) needed by patients on the first 24 hours after spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hermann dos Santos Fernandes, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, if requested
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publishing the study. No time limit.
Access Criteria: If requested

REFERENCES:
- [Background] Anger M, Valovska T, Beloeil H, Lirk P, Joshi GP, Van de Velde M, Raeder J; PROSPECT Working Group* and the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guideline for total hip arthroplasty: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Aug;76(8):1082-1097. doi: 10.1111/anae.15498. Epub 2021 May 20. PMID 34015859
- [Background] Panzenbeck P, von Keudell A, Joshi GP, Xu CX, Vlassakov K, Schreiber KL, Rathmell JP, Lirk P. Procedure-specific acute pain trajectory after elective total hip arthroplasty: systematic review and data synthesis. Br J Anaesth. 2021 Jul;127(1):110-132. doi: 10.1016/j.bja.2021.02.036. PMID 34147158
- [Background] Li D, Yang Z, Xie X, Zhao J, Kang P. Adductor canal block provides better performance after total knee arthroplasty compared with femoral nerve block: a systematic review and meta-analysis. Int Orthop. 2016 May;40(5):925-33. doi: 10.1007/s00264-015-2998-x. Epub 2015 Oct 10. PMID 26452678
- [Background] Bugada D, Bellini V, Lorini LF, Mariano ER. Update on Selective Regional Analgesia for Hip Surgery Patients. Anesthesiol Clin. 2018 Sep;36(3):403-415. doi: 10.1016/j.anclin.2018.04.001. Epub 2018 Jul 11. PMID 30092937
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667